CLINICAL TRIAL: NCT03423979
Title: Evaluation of Optilume™ BPH Prostatic Drug Coated Balloon Dilation Catheter in the Treatment of Moderate-to-Severe Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia
Brief Title: Optilume™ BPH Prostatic Drug Coated Balloon Dilation Catheter
Acronym: EVEREST-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR1051
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: treatment group - treated with Optilume™ BPH Prostatic Drug Coated Balloon Dilation Catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Optilume™ BPH Prostatic DCB Dilation Catheter (Experimental): Optilume™ BPH Prostatic DCB treatment procedure
  Interventions: Device: Optilume™ BPH Prostatic DCB Dilation Catheter; Drug: Paclitaxel

INTERVENTIONS:
Device: Optilume™ BPH Prostatic DCB Dilation Catheter — BPH Prostatic DCB treatment - The Optilume BPH Prostatic DCB Dilation Catheter System should be prepared per the Instructions for Use (IFU).
  Other Names: BPH Prostatic DCB
Drug: Paclitaxel — paclitaxel will release to adjacent tissue after the balloon inflated in the urethra
  Other Names: drug coated balloon

SUMMARY:
A prospective, non-randomized study. The subjects will be enrolled and treated with the Optilume BPH Prostatic DCB Dilation Catheter System at up to 8 clinical sites. The post-treatment follow-up visit can be up to 5 years.

The objective of the study is to evaluate the safety and efficacy of the Optilume™ BPH Prostatic Drug Coated Balloon Dilation Catheter System in the treatment of BPH.

DETAILED DESCRIPTION:
A prospective, non-randomized, multi-center study. The study will enroll up to 85 subjects to be enrolled and treated with the Optilume BPH Prostatic DCB Dilation Catheter System at up to 8 clinical sites. Subjects will be followed up post-treatment at Foley removal, and up to 1 year. The subjects may choose to be followed-up annually for 5 years or until study close, whichever comes first.

Study device is Optilume™ BPH Prostatic Drug Coated Balloon Dilation Catheter System.

Study primarily outcomes are measured by 1). Change in IPSS score at 3-month post-procedure follow-up; 2). Major device or procedure related complications at 3-month post-procedure follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject > 50 years of age who has moderate-to-severe LUTS (IPSS score of ≥ 13) and is a candidate for interventional therapy
2. LUTS felt to be secondary to an enlarged prostate (henceforth termed LUTS/BPH)
3. Peak urinary flow rate (Qmax) ≥ 5 mL/sec and ≤ 15 ml/sec with minimum voided volume of ≥ 125 ml
4. Post-void residual (PVR) ≤ 250 ml
5. Prostate volume 20 - 80 gm as determined by TRUS
6. Prostatic urethra length is 35 - 55 mm as determined by TRUS
7. Able to complete the study protocol in the opinion of the investigator

Exclusion Criteria:

1. Interested in maintaining fertility and unwilling to use protected sex for the first 30 days post treatment
2. Unwilling to abstain or use protected sex for ninety (90) days post treatment if sexual partner is of child bearing potential
3. Presence of a penile implant or stent(s) in the urethra or prostate
4. Any prior minimally invasive intervention (e.g. TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
5. PSA > 10 ng/ml unless prostate cancer is ruled out by biopsy. If PSA is > 4 ng/ml and ≤ 10 ng/ml, prostate cancer must be ruled out to the satisfaction of the investigator via additional tests including digital rectal exam (DRE) and/or biopsy
6. Confirmed or suspected malignancy of prostate or bladder
7. Active or history of epididymitis within the past 3 months
8. Previous pelvic irradiation or radical pelvic surgery
9. Documented active urinary tract infection (UTI) by culture or bacterial prostatitis within last year documented by culture (UTI is defined as >100,000 colonies per ml urine from midstream clean catch or catheterization specimen)
10. Visible hematuria with subject urine sample without known contributing factor
11. Neurogenic bladder or sphincter abnormalities or neurological disorders that might affect bladder or sphincter function
12. Previous or current diagnosis of urethral strictures, bladder neck contracture or detrusor muscle spasms
13. Use of beta blockers, antihistamines, anticonvulsants, or antispasmodics within 1 week prior to treatment unless there is documented evidence of stable dosing for last 6 months (no dose changes)
14. Use of alpha blockers, antidepressants, anticholinergics, androgens, daily tadalafil or gonadotropin-releasing hormonal analogs (prescribed for BPH) within 3 weeks prior to treatment
15. Use of 5-alpha reductase inhibitor within 6 months prior to treatment
16. Incidence of spontaneous urinary retention within 6 months prior to baseline assessment
17. Post-void residual volume > 250 ml or catheter dependent bladder drainage
18. Overactive bladder (OAB) or urge incontinence
19. Known poor detrusor muscle function (e.g. Qmax < 5 ml/sec)
20. Current bladder stones or prostatic calculi
21. Biopsy of prostate within 30 days prior to procedure or planned within 30 days following the procedure
22. History of cancer in non-genitourinary system which is not considered cured (except basal cell or squamous cell carcinoma of the skin). A potential participant is considered cured if there has been no evidence of cancer within five years
23. History of clinically significant comorbidities or presence of unstable conditions (e.g. cardiovascular, lung, renal [serum creatinine > 2.0 mg/dl], hepatic, bleeding disorders, or metabolic impairment) that may confound the results of the study or have a risk to subject per investigator's opinion
24. Any cognitive disorder that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affects the ability to complete the study quality of life questionnaires
25. Expected life expectancy < one year
26. Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with all the follow-up requirements
27. Currently enrolled in or plan to enroll in another investigational clinical trial for any disease except for observational only study
28. In the opinion of the investigator, it is not in the subject's best interest to participate in the study
29. Current treatment with anti-coagulants (e.g., warfarin or enoxaparin) or anti-platelet medications other than aspirin (e.g., clopidogrel)
30. Anatomy, e.g. presence of false passage or size of meatus, is not suitable for treatment in this study
31. Device that corresponds with the subject's prostate size per the IFU is not available
32. Intravesical prostatic protrusion (IPP) > 1 cm
33. Current uncontrolled diabetes (hemoglobin A1c > 7%)
34. Unable or unwilling to provide all the protocol-required semen samples
35. Sensitivity to paclitaxel, on medication that may have negative interaction with paclitaxel, or contraindicated for systemic paclitaxel

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on biological sex
Enrollment: 80 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2024-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Moland, Study Director — Urotronic Inc.
Locations (5):
- Dominican Republic (3):
  - Union Medica Hospital, Santiago de los Caballeros, Santiago Province
  - Urolaser SRL, Santo Domingo Oeste, Santo Domingo Province
  - Centro Medico Dr. Canela, SRL, La Romana
- Panama (2):
  - Consultorios Royal Center, Panama City, Urbanización Marbella Ciudad de Panamá
  - Centro Especializado San Fernando, Panama City

REFERENCES:
- [Derived] Pichardo M, Rijo E, Espino G, Lay RR, Estrella R, Gonzalez C, Fernandez M, Soriano D, Peralta IM, Kaplan SA. Durable benefit after treatment of obstructive benign prostatic hyperplasia with a novel drug-device combination product: 2-year outcomes from the EVEREST-I study. World J Urol. 2023 Aug;41(8):2209-2215. doi: 10.1007/s00345-023-04473-1. Epub 2023 Jun 24. PMID 37354260

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optilume™ BPH Prostatic DCB Dilation Catheter
Started | 80
Completed | 52
Not Completed | 28
Not completed — Death | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Arm/Group | Optilume™ BPH Prostatic DCB Dilation Catheter
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black/African Origin | 10
  Race/Ethnicity: Caucasian | 2
  Race/Ethnicity: Hispanic/Latino | 68
Prostate Volume (g) [Mean (Standard Deviation); unit: grams] | 35.9 (13.2)
Presence of Intravesical Prostatic Protrusion [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Responder at 3 Months
Description: The proportion of subjects experiencing at least a 40% improvement in International Prostate Symptom Score (IPSS) scores from baseline to 3 months. The IPSS contains the well-validated, highly reliable and responsive American Urological Association symptom score (AUASS) assessment to identify the severity of BPH symptoms. The first seven questions in the IPSS address frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying, and urgency, and scored on a 6-point scale (0 to 5). The IPSS can be interpreted as follows: 0-7 mildly symptomatic, 8-19 moderately symptomatic, and 20-35 severely symptomatic.
Time Frame: 90 days
Population: In the primary analysis, a worst-case approach was used where those missing 3 month IPSS scores were imputed as non-responders
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume™ BPH Prostatic DCB Dilation Catheter
Number analyzed (Participants) | 80
Participants | 65

2. Primary Outcome: Major Device/Procedure Related Complications
Description: The proportion of subjects reporting a composite of device/procedure related severe urinary retention (lasting >14 days), unresolved stress urinary incontinence, or bleeding requiring transfusion.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Optilume™ BPH Prostatic DCB Dilation Catheter
Number analyzed (Participants) | 80
Participants | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Optilume™ BPH Prostatic DCB Dilation Catheter
All-Cause Mortality (participants affected / at risk) | 5/80
Serious Adverse Events (participants affected / at risk) | 25/80
Other Adverse Events (participants affected / at risk) | 50/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optilume™ BPH Prostatic DCB Dilation Catheter (N=80)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 8 (8)
Urethral Stenosis (Renal and urinary disorders) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 3 (3)
Anesthetic Complication (Pulmonary) (Injury, poisoning and procedural complications) | 1 (1)
Complication of Device Removal (General disorders) | 2 (2)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Urethral Perforation (Renal and urinary disorders) | 1 (1)
Rectal Perforation (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Death related to heart failure/Thrombosis (Vascular disorders) | 1 (1)
High Blood Pressure (Vascular disorders) | 1 (1)
Oral lesion (cancer) (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optilume™ BPH Prostatic DCB Dilation Catheter (N=80)
Hematuria (Renal and urinary disorders) | 15 (15)
Urinary Retention (Renal and urinary disorders) | 9 (10)
Urinary Incontinence (Renal and urinary disorders) | 11 (13)
Dysuria (Renal and urinary disorders) | 10 (10)
Ejaculation Disorder (Reproductive system and breast disorders) | 8 (8)
Urinary Tract Infection (Infections and infestations) | 14 (15)

LIMITATIONS AND CAVEATS:
Interim review of safety data lead to refinement of device sizing and appropriate device size selection based on prostate dimensions for the final 30 subjects enrolled. Safety information reported for full cohort, as no pre-specified sub-analyses were planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT03423979/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03423979/SAP_002.pdf